CLINICAL TRIAL: NCT00739024
Title: A Randomized, Double-blind Placebo-controlled, Parallel Group Study to Study the Efficacy and Tolerability of Ramelteon (Rozerem) in the Prophylaxis of Migraine
Brief Title: A Study of a Melatonin Receptor Agonist to Prevent Migraine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment slow and administrative reasons
Sponsor: Swedish Medical Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRC 0690
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura
Keywords: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Active Comparator): Ramelteon once daily (double-blind assignment)
  Interventions: Drug: Ramelteon
- Placebo (Placebo Comparator): Placebo tablet, once daily (double-blind assignment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — 8 mg tablet, oral, once daily
  Other Names: Rozerem
  Arms: Active Treatment
Drug: Placebo — Placebo tablet, oral, once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if ramelteon will reduce the number of migraine headaches over a 12 week period. The safety and tolerability of ramelteon will also be evaluated. Ramelteon has been approved by the U.S. Food and Drug Administration (FDA) for insomnia (trouble sleeping); however; ramelteon has not been approved for the prevention of migraines.

DETAILED DESCRIPTION:
Sleep has played an important role in migraine. Younger migraine sufferers usually report relief of migraine after sleep. In older migraine sufferers migraine is sometimes triggered with sleep changes. Occurrence of migraine in the early morning is very common. Therefore in these individuals regulation of sleep may improve the frequency of migraine. Recent PET studies done during migraine demonstrated activation of hypothalamus during migraine. In light of this new data and the known action of ramelteon on the melatonin receptors it may theoretically provide an insight on a possible mechanism of action in migraine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18 to 65 years, inclusive.
* An established history of migraine, with or without aura and probable migraine, conforming to the revised IHS criteria (2004) for at least 1 year before screening, sufficient to establish the diagnosis.
* To be randomized, during the prospective 4-week baseline period (approximately 28 days before Visit 2), subjects must have more than 4 migraine/probable migraine attacks per month (using the 24-hour rule).
* Must have been less than 50 years of age at the time of initial migraine onset.
* Must have no clinically significant and relevant abnormalities on physical or neurologic examinations
* Must have completed a washout of all prophylactic medications for migraine before the start of the 4-week prospective baseline period (ie, 28 days before Visit 2, when randomization occurs).
* Female subjects must be at least 1 of the following:
* postmenopausal, or
* surgically incapable of being children, or
* practicing a highly effective method of birth control

Exclusion Criteria:

* Most frequent type of headache does not meet the revised IHS diagnostic criteria for migraine with aura or without aura or probable migraine.
* Pregnant or lactating women, or sexually active women of childbearing potential who are not using an appropriate method of contraception.
* Failed adequate trials of prophylactic agents with demonstrated or possible efficacy in the prophylaxis of migraine. These agents include beta-blockers, tricyclic antidepressants, valproate, topiramate, and methysergide.
* Unable to complete the diary in a timely and accurate manner after each migraine headache attacks, either independently or with assistance.
* Overuse of analgesics or specific agents for abortive treatment of migraine attacks, which makes the investigator suspect medication overuse headache.
* Receiving non-pharmacological prophylactic treatments such as acupuncture, chiropractic, or massage, if these were started less than 1 month before the screening visit (Day -28). These therapies may be continued if started before that time.
* Currently abusing alcohol or other drugs.
* Have a central nervous system neoplasm or infection, demyelinating disease, degenerative or progressive central nervous system disease, or active epilepsy.
* History of serious systemic disease, including hepatic insufficiency, renal insufficiency, a malignant neoplasm, any disorder in which prognosis for survival is less than 3 months, or any disorder which in the judgment of the investigator will place the subject at excessive risk by participation in a controlled trial.
* Have a significant psychiatric disorder, such as acute psychosis, schizophrenia, severe bipolar disorder, or severe unipolar mood disorder, of sufficient severity to preclude safe and effective participation of the subject in the study.
* Require continued use of any of protocol-defined prohibited medications during the study
* Have any recent or remote history of suicide attempt or ideation
* Known or strongly suspected to be non-compliant in administering daily medications.
* Received an experimental drug or used an experimental device within 30 days before the Screening Visit.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator
* Any reason for which the investigator, upon her evaluation, feels that it is in the subject's best interest not to continue on in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheena K Aurora, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Pain and Headache Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8/2008 through March 2010, clinic setting
Pre-assignment Details: 18 Participants signed Informed Consent. 5 did not qualify for randomization. 13 participants were randomized to Active Treatment or Placebo.
Groups:
- Active Treatment: Random assignment to active treatment
- Placebo: Random assignment to placebo
Period: Overall Study
Arm/Group | Active Treatment | Placebo
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: T-Test
Description: It was planned to use a simple T-Test or ANoVa for data analysis. No Analysis was made due to insufficient recruitment. Planned primary efficacy variable was the percent reduction in the average monthly miqraine/probable migraine frequency from the baseline period to the entire double-blind treatment phase of the study.
Time Frame: 4 weeks
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Active Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No